CLINICAL TRIAL: NCT07006935
Title: Pilot Study of the Cognitive and Neurobiological Effects of the Clubhouse Model of Psychosocial Rehabilitation for Schizophrenia and Related Conditions
Brief Title: REACH Study (Recovery Environments: Assessing Cognitive & Brain Health in Community Mental Health)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Magnolia Clubhouse (Unknown); The Centers (Unknown)
Responsible Party: Principal Investigator, Jessica Wojtalik, Assistant Professor, Case Western Reserve University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20250623
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia; Schizo Affective Disorder; Schizophreniform Disorders
Keywords: Clubhouse Model of Psychosocial Rehabilitation; Community mental health interventions; Cognition; Brain functioning
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clubhouse Model of Psychosocial Rehabilitation for Serious Mental Illness (Experimental): The Clubhouse Model (CM) is a strengths-focused, evidence-based, and comprehensive approach to psychosocial rehabilitation for serious mental illness. The CM uses an intentional community of support to create a safe and holistic setting to practice real-world functioning. The core of the CM is the 'work-ordered day,' a concept where members, as opposed to patients, are integral to and needed for the successful daily operation of the Clubhouse. Members choose a 'work unit' each day of attendance. Most clubhouses have four work units, such as (1) Administration (e.g., database management); (2) Hospitality (e.g., Clubhouse cafe); (3) Membership (e.g., employment programs); and (4) Communications (e.g., newsletter). Other unique aspects include its voluntary and humanistic nature, prioritization of member choice, unrestricted and flexible membership, and the elimination of provider-patient hierarchy. The CM has a sophisticated accreditation process based on 37 international standards.
  Interventions: Behavioral: Clubhouse Model of Psychosocial Rehabilitation for Serious Mental Illness
- Usual Community-Based Mental Health Care (Active Comparator): Usual care includes services typically available in the community at mental health agencies, including case management, Assertive Community Treatment, counseling, peer support services, psychoeducational support groups, family support groups, supported education/employment, permanent supportive housing, and medication management.
  Interventions: Behavioral: Usual Community-Based Mental Health Care

INTERVENTIONS:
Behavioral: Clubhouse Model of Psychosocial Rehabilitation for Serious Mental Illness — The Clubhouse Model (CM) is a strengths-focused, evidence-based, and comprehensive approach to psychosocial rehabilitation for serious mental illness. The CM uses an intentional community of support to create a safe and holistic setting to practice real-world functioning. The core of the CM is the 'work-ordered day,' a concept where members, as opposed to patients, are integral to and needed for the successful daily operation of the Clubhouse. Members choose a 'work unit' each day of attendance. Most clubhouses have four work units, such as (1) Administration (e.g., database management); (2) Hospitality (e.g., Clubhouse cafe); (3) Membership (e.g., employment programs); and (4) Communications (e.g., newsletter). Other unique aspects include its voluntary and humanistic nature, prioritization of member choice, unrestricted and flexible membership, and the elimination of provider-patient hierarchy. The CM has a sophisticated accreditation process based on 37 international standards.
  Arms: Clubhouse Model of Psychosocial Rehabilitation for Serious Mental Illness
Behavioral: Usual Community-Based Mental Health Care — Usual care includes services typically available in the community at mental health agencies, including case management, Assertive Community Treatment, counseling, peer support services, psychoeducational support groups, family support groups, supported education/employment, permanent supportive housing, and medication management.
  Arms: Usual Community-Based Mental Health Care

SUMMARY:
The purpose of this study is to understand how different types of community-based mental health care affect thinking abilities, daily functioning, and brain activity in adults with schizophrenia and related conditions. The investigators are especially interested in learning whether the Clubhouse Model-a structured, supportive community for individuals with mental illness-has unique benefits compared to standard outpatient mental health services. If participants decide to join, they will be asked to complete a total of six study visits with the research team over the course of your participation. Three of these study visits are at the beginning (baseline) and the remaining three are six months later. Two of the three visits will includes interviews, questionnaires, and thinking and memory tasks (cognitive testing) and one session will be an MRI brain scan, which is a safe and non-invasive imaging procedure. The total time required for each visit will be approximately 90 minutes to two hours. Participants may take breaks as needed.

ELIGIBILITY:
Inclusion Criteria:

* (1) have a DSM-V diagnosis of schizophrenia, schizoaffective disorder, or schizophreniform confirmed by diagnostic assessment and medical record review
* (2) between the ages of 18-50
* (3) stabilized on psychotropic medication as indicated by no changes to the primary psychiatric medication in the last month
* (4) able to read and speak fluent English at a sixth grade level or higher for purposes of informed consent and cognitive testing
* For Clubhouse members, they must be a first-time, newly enrolled member

Exclusion Criteria:

* (1) had previous membership at a Clubhouse (Magnolia or elsewhere)
* (2) have a current severe substance use disorder
* (3) have persistent suicidal or homicidal behavior
* (4) a co-occurring diagnosis of an intellectual or learning disability or neurodevelopment condition (e.g., Autism; based on chart review)
* (5) had recent psychiatric instability requiring hospitalization in the past month;
* (6) history of a traumatic brain injury (TBI; based on record review)
* (7) contraindicators for MRI (e.g., pacemaker, claustrophobia)
* Participants in the usual care will be excluded if they are a current Clubhouse member or join a Clubhouse during participation in this research

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in overall cognitive performance as measured by MATRICS Consensus Cognitive Battery (MCCB) | Baseline and 6 months
  The MATRICS Consensus Cognitive Battery (MCCB), which was developed by NIMH as a standardized assessment tool as an outcome measure of cognitive change in intervention trials. This performance-based battery contains 10 field standard, individually administered computer and paper-and-pencil tests of neurocognition (processing speed, attention, working memory, verbal learning, visual learning, and problem solving) and social cognition. The MCCB takes approximately 60-90 minutes to administer. The overall composite score (M = 50, SD = 10) with higher scores indicated better cognitive performance.
Change in functional outcome as measured by Specific Levels of Functioning Scale (SLOF) | Baseline and 6 months
  The SLOF is a 30-item self-and/or informant-report measure of interpersonal relationships, social acceptability, community activities, and living and work skills rated on a 5-point scale, with higher scores reflecting better functional outcome.
Change in quality of life as measured by World Health Organization Quality of Life Brief Assessment (WHOQOL-BREF) | Baseline and 6 months
  The WHOQOL-BREF is a 26-item quality of life (QoL) measure developed by the World Health Organization of physical health, psychological, social relationships, and environment QoL. Items are rated on a 5-point scale, with higher scores reflecting better QoL.
Change in disability as measured by the 12-item WHO Disability Assessment Schedule 2.0 (WHODAS 2.0 | Baseline and 6 months
  A brief (12-item), universal interviewer/self-report measure of functional disability that assesses 6 areas (mobility, life activities, cognition, participation, self-care, getting along with others) rated on level of difficulty in the past 30 days with higher scores indicating more disability.
Change in task-based brain activation during functional MRI (fMRI) as measured by the AX-Continuous Performance Task (AX-CPT) | Baseline and 6 months
  An NIMH validated fMRI task of goal maintenance (attention) in schizophrenia. This task implements the "A-then-X rule" where participants are instructed to make an index finger button press only when "A" precedes "X" (target trial, 72%) and a middle finger press for all other "non-target" trials (AY: 11%; BX: 11%; BY: 6%) for a total of 4 blocks of 36 trials (144 total). Trials are presented for 500ms followed by a cue (+) presentation for 1000ms (target or non-target response expected) with an interstimulus interval of 2000ms. Instructions and practice trials are embedded. The main contrast of interest for group-level analyses is the high vs. low cognitive load trials (cue A > cue B), with greater fronto-limbic brain activation during high cognitive load indicating strong attention-related brain activation.
Change in task-based brain activation during functional MRI (fMRI) as measured by the Emotional Faces N-Based Task (EFNBACK) | Baseline and 6 months
  A modified version of the standard working memory n-back task. This task includes 8 blocks (4 are 0-back and 4 are 2-back) of 12 trials. Each block starts with instructions indicating the condition (0-back or 2-back) presented for 3500ms, which is followed by the target stimulus (letters) flanked by emotional valence distractor conditions (happy, fearful, neutral, or no face) for 500ms, with an interstimulus interval jittered at an average of 3500ms. Blocks with emotional vs. no distractors are randomly interspersed throughout. The main contrasts of interest for group-level analyses are working memory load (2-back > 0-back) and emotion distractor conditions (happy > neutral; fearful > neutral), with greater activation during the 2-back and emotional distractor conditions indicating better working memory and emotion regulation brain functioning.

SECONDARY OUTCOMES:
Change in social cognition (emotion recognition) as measured by Penn Emotion Recognition Task (ER-40) | Baseline and 6 months
  Measures the ability to accurately identify different emotions (i.e., happy, sad, anger, and fear) in 40 colored images of human faces with a computer-administered, performance-based, and forced-choice format. Generates a total score of correctly identified emotions, with higher scores indicative of better emotional recognition ability.
Change in social cognition (social inference) as measured by The Awareness of Social Inference Test, part III (TASIT) | Baseline and 6 months
  The TASIT is a performance-based assessment that includes 16 short video vignettes (15 to 60 seconds) of social exchanges between actors. After watching a vignette, participants are asked four questions regarding their perceptions of lies or sarcasm in the social exchange. A total score is generated of correct responses, with higher scores indicative of better social inference ability.
Change in social cognition (theory of mind) as measured by the Hinting Task | Baseline and 6 months
  Requires theory of mind to infer the genuine intentions of a character's indirect speech to a second character across 10 short stories read by the test administrator. Created as a performance-based measure of theory of mind ability in people with schizophrenia. A total score of correct responses is yielded, with higher scores reflecting stronger ability to correctly perceive the hint of the character's true intention.
Change in functional capacity as measured by he UCSD Performance-Based Skills Assessment, Brief version (UPSA-B) | Baseline and 6 months
  The UCSD Performance-Based Skills Assessment is a brief performance-based measure of functional capacity of financial and communication skills. Scores range from 0 to 100, with higher scores indicating better functional capacity.
Change in Self-Efficacy as measured by the New General Self-Efficacy Scale (NGSE) | Baseline and 6 months
  The New General Self-Efficacy Scale (NGSE) is an 8-item self-report questionnaire designed to assess an individual's overall belief in their ability to perform well across a variety of situations. Respondents rate their agreement with each statement on a 5-point Likert scale, ranging from 0 (strongly disagree) to 4 (strongly agree). The total score range is from 0-32 with higher scores indicating greater self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A Wojtalik, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No